CLINICAL TRIAL: NCT02189694
Title: An Open-label, Randomized, Three-way, Cross-over Study to Assess the Efficacy of Single-hormone Closed-loop Strategy, Dual-hormone Closed-loop Strategy and Conventional Pump Therapy in Regulating Overnight Glucose Levels in Children With Type 1 Diabetes in a Diabetes Camp
Brief Title: Closed-loop Control of Overnight Glucose Levels (Artificial Pancreas) in Children With Type 1 Diabetes in a Diabetes Camp
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Collaborators: Montreal Children's Hospital of the MUHC (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Associate professor of Medicine, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLASS-08
Record Dates: First submitted 2014-07-03; First posted 2014-07-14 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Hypoglycemia; Insulin; Glucagon; Closed-loop system; Artificial pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Insulin pump therapy (Active Comparator): Glucose levels will be controlled for 3 consecutive nights using insulin pump therapy. Subjects will carry on with their normal conventional insulin pump therapy and will be allowed to freely implement therapeutic adjustments..
  Interventions: Device: Insulin pump therapy
- Single-hormone closed-loop strategy (Active Comparator): Glucose levels will be controlled by single-hormone closed-loop strategy for 3 consecutive nights. A member of the research team will be present at the diabetic camp to ensure protocol implementation and patient's safety. Glucose levels will be controlled by single-hormone closed-loop strategy between 22:00 until 7:00 next morning. Glucose sensor reading will be entered manually into the computer every 10 minutes. The computer will generate a recommendation for the basal rates of insulin delivery. Pump's parameters will then be changed manually to implement the computer generated recommendations.
  Interventions: Device: Single-hormone closed-loop strategy
- Dual-hormone closed-loop strategy (Active Comparator): Glucose levels will be controlled by dual-hormone closed-loop strategy for 3 consecutive nights. A member of the research team will be present at the diabetic camp to ensure protocol implementation and patient's safety. Glucose levels will be controlled by dual-hormone closed-loop strategy between 22:00 until 7:00 next morning. Glucose sensor readings will be entered manually into the computer every 10 minutes. The computer will generate a recommendation for the basal rates of insulin delivery and glucagon mini-boluses. Pumps' parameters will then be changed manually to implement the computer generated recommendations.
  Interventions: Device: Dual-hormone closed-loop strategy

INTERVENTIONS:
Device: Single-hormone closed-loop strategy — Variable subcutaneous insulin infusion rates will be used to regulate glucose levels. Insulin Aspart (Novorapid, Novo Nordisk) will be used.
  Arms: Single-hormone closed-loop strategy
Device: Dual-hormone closed-loop strategy — Variable subcutaneous insulin and glucagon infusion rates will be used to regulate glucose levels. Insulin Aspart (Novorapid, Novo Nordisk) and Glucagon (Eli Lilly and Company) will be used.
  Arms: Dual-hormone closed-loop strategy
Device: Insulin pump therapy — Subjects will use conventional pump therapy to regulate glucose levels. Insulin Aspart (Novorapid, Novo Nordisk) will be used.
  Arms: Insulin pump therapy

SUMMARY:
Closed-loop strategy is composed of three components: glucose sensor to read glucose levels, insulin pump to infuse insulin and a dosing mathematical algorithm to decide on the required insulin dosages based on the sensor's readings. A dual-hormone closed-loop system would regulate glucose levels through the infusion of two hormone: insulin and glucagon.

The main objective of this project is to compare the efficacy of single-hormone closed-loop strategy, dual-hormone closed-loop strategy and pump therapy to regulate overnight glucose levels in children with type 1 diabetes in a diabetes camp.

The investigators hypothesized that dual-hormone closed-loop strategy reduces the time spent in hypoglycemia in children with type 1 diabetes (T1D) compared to single-hormone closed-loop strategy, which in turn is more effective than the conventional pump therapy to reduce time spent in hypoglycemia

DETAILED DESCRIPTION:
Closed-loop strategy is composed of three components: glucose sensor to read glucose levels, insulin pump to infuse insulin and a dosing mathematical algorithm to decide on the required insulin dosages based on the sensor's readings. A dual-hormone closed-loop system would regulate glucose levels through the infusion of two hormone: insulin and glucagon.

The investigators aim to conduct a randomized three-way cross-over trial comparing single hormone closed-loop strategy, dual-hormone closed-loop strategy and the conventional pump therapy. The investigators aim to compare the three interventions for 3 consecutive nights in children with type 1 diabetes in a diabetes camp.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between the 8 and 17 years of old.
* Clinical diagnosis of type 1 diabetes for at least one year. The subject will have been on insulin pump therapy for at least 3 months.
* HbA1c ≤ 11.0%.

Exclusion Criteria:

* Clinically significant nephropathy, neuropathy or retinopathy as judged by the investigator.
* Severe hypoglycemic episode within two weeks of inclusion in the study. A severe hypoglycemic episode is defined as loss of conscience, seizure or a hospital emergency visit.
* Current use of oral glucocorticoid medication (except low stable dose according to investigator judgement). Stable doses of inhaled steroids are acceptable.
* Known or suspected allergy to the trial products.
* Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator.
* Failure to comply with team's recommendations (e.g. not willing to use trial pump, etc).

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Percentage of time of glucose levels spent below 4.0 mmol/L. | Up to 8 hours

SECONDARY OUTCOMES:
Percentage of time of glucose levels spent between 4.0 and 8.0 mmol/L | Up to 8 hours
Percentage of time of glucose levels spent below 3.5 mmol/L | Up to 8 hours
Percentage of time of glucose levels spent below 3.3 mmol/L | Up to 8 hours
Percentage of time of glucose levels spent above 8 mmol/L | Up to 8 hours
Percentage of time of glucose levels spent above 10 mmol/L. | Up to 8 hours
Area under the curve of glucose levels below 4.0 mmol/L | Up to 8 hours
Area under the curve of glucose levels below 3.5 mmol/L | Up to 8 hours
Area under the curve of glucose levels below 3.3 mmol/L | Up to 8 hours
Area under the curve of glucose levels above 8.0 mmol/L | Up to 8 hours
Area under the curve of glucose levels above 10.0 mmol/L. | Up to 8 hours
Mean glucose levels. | Up to 8 hours
Standard deviation of glucose levels | Up to 8 hours
  Measure of glucose variability.
Total insulin delivery | Up to 8 hours
Hypoglycemic risk assessed by the total number of hypoglycemic event (> 15 minutes) below 3.1 mmol/L | Up to 8 hours
Hypoglycemic risk assessed by the number of patients experiencing at least one hypoglycemic event (> 15 minutes) below 3.1 mmol/L | Up to 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, MD, PhD, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Haidar A, Legault L, Matteau-Pelletier L, Messier V, Dallaire M, Ladouceur M, Rabasa-Lhoret R. Outpatient overnight glucose control with dual-hormone artificial pancreas, single-hormone artificial pancreas, or conventional insulin pump therapy in children and adolescents with type 1 diabetes: an open-label, randomised controlled trial. Lancet Diabetes Endocrinol. 2015 Aug;3(8):595-604. doi: 10.1016/S2213-8587(15)00141-2. Epub 2015 Jun 8. PMID 26066705